CLINICAL TRIAL: NCT01324453
Title: Phase II Clinical Trial to Evaluate the Benefits of Postconditioning in STEMI
Brief Title: Phase II Clinical Trial to Evaluate the Benefits of Postconditioning in ST-Elevation Myocardial Infarction (STEMI)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: opt004; 1R01HL103927-01A1 (NIH)
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; STEMI; Post Conditioning; Primary Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post conditioning + PCI (Experimental)
  Interventions: Procedure: Post Conditioning + Primary PCI
- Standard PCI (Active Comparator)
  Interventions: Procedure: Standard Primary PCI

INTERVENTIONS:
Procedure: Post Conditioning + Primary PCI — Four, 30-second PTCA balloon occlusions followed by 30-seconds of reperfusion over a total of 4 minutes, in addition to Percutaneous Coronary Intervention as clinically indicated.
  Arms: Post conditioning + PCI
Procedure: Standard Primary PCI — Routine Percutaneous Coronary Intervention as clinically indicated.
  Arms: Standard PCI

SUMMARY:
This study will evaluate change in heart muscle function from baseline to three months and twelve months in participants who present with a heart attack and a completely occluded coronary artery. These subjects will be randomized to receive standard Percutaneous transluminal coronary angioplasty (PTCA)/Stenting to open the artery or routine PTCA/Stenting plus post conditioning. Post conditioning commences immediately upon reperfusion using four cycles of thirty second inflations with a standard angioplasty balloon followed by a thirty seconds of reperfusion. The investigators hypothesize that Postconditioning reduces the size of the heart attack when utilized with successful primary Angioplasty/stent.

DETAILED DESCRIPTION:
Single center study involving 140 patients randomized to Post Conditioning + Percutaneous coronary intervention (PCI) versus routine PCI during their ST-Elevation Myocardial Infarction (STEMI, Heart Attack) presentation. The Post Conditioning protocol consists of performing four, 30-second PTCA (Angioplasty) balloon occlusions followed by 30-seconds of reperfusion over a total of 4 minutes. The first balloon inflation occurs immediately after an angioplasty guidewire is placed through the obstruction in the artery. Following this protocol the vessel is stented as part of the usual practice for treatment of STEMI. No other treatment differences will occur between the two groups and all patients will receive the usual post-STEMI care. Patients in both groups will receive a cardiac MRI 3-5 days following their STEMI for measurement of heart attack size and heart muscle function, among other measures. Patients will undergo collection of blood for creatine kinase (CK)-MB and troponin I every 8 hours for 24 hours following PCI. All patients will be followed by phone follow-up visits to review history and major adverse cardiac event (MACE) (death, recurrent STEMI, repeat revascularization, arrhythmias, implantable cardioverter-defibrillator (ICD) placement and hospitalization for congestive heart failure (CHF)). All patients will be required to take P2Y12 inhibitors and aspirin for the duration of the trial. All patients will be treated with angiotensin-converting enzyme inhibitor (ACE-I), beta blockers and statins.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old, < 80 years old
* Able to give informed consent
* Able to undergo cMRl (cardiac magnetic resonance imaging
* ST-segment elevation infarction with 100% occlusion of a major epicardial vessel (> 2.5 mm)
* No angiographic evidence of collateral flow distal to occluded artery
* Ischemic duration between 1.0 and 6 hours
* Thrombolysis in myocardial infarction (TIMI) 3 Flow following PCI

Exclusion Criteria:

* Visible collateral blood flow to the distal vasculature of the occluded vessel
* Previous Coronary Artery Bypass Graft surgery
* Previous q-wave myocardial infarction in the same territory
* Inability to give informed consent
* Inability to undergo cMRl
* Life expectancy less than one year
* History of Non-compliance or alcohol or drug addiction
* Patients with cardiogenic shock, cardiac arrest, hypothermia on presentation
* Chronic dialysis or significant renal insufficiency (Creatinine Clearance < 35 mI/mm/i .73 m2)
* TIMI Flow > 0 on presentation
* Ischemic Time > 6 hours or < 1.0 hours
* Presence of significant valvular heart disease (>mod Aortic Stenosis, >2+ Mitral Regurgitation)
* Known Left Ventricular systolic dysfunction (Left Ventricular Ejection Fraction < 50% prior to STEMI)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-03; Primary Completion 2016-11 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay H Traverse, MD, Principal Investigator — Minneapolis Heart Institute Foundation at Abbott Northwestern Hospital
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Traverse JH, Swingen CM, Henry TD, Fox J, Wang YL, Chavez IJ, Lips DL, Lesser JR, Pedersen WR, Burke NM, Pai A, Lindberg JL, Garberich RF. NHLBI-Sponsored Randomized Trial of Postconditioning During Primary Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction. Circ Res. 2019 Mar;124(5):769-778. doi: 10.1161/CIRCRESAHA.118.314060. PMID 30602360

RESULTS

PARTICIPANT FLOW:
Groups:
- Post Conditioning + Percutaneous Coronary Intervertion (PCI): Post Conditioning + Primary PCI: Four, 30-second percutaneous transluminal coronary angioplasty (PTCA) balloon occlusions followed by 30-seconds of reperfusion over a total of 4 minutes, in addition to PCI as clinically indicated.
- Standard Percutaneous Coronary Internvention (PCI): Standard Primary PCI: Routine Percutaneous Coronary Intervention as clinically indicated.
Period: Overall Study
Arm/Group | Post Conditioning + Percutaneous Coronary Intervertion (PCI) | Standard Percutaneous Coronary Internvention (PCI)
Started | 54 | 49
Completed | 54 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post Conditioning + PCI | Standard PCI | Total
Number analyzed (Participants) | 54 | 49 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (10.0) | 60.0 (9.7) | 59.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 48 | 39 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 48 | 46 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Diabetes [Count of Participants; unit: Participants]
  Diabetes | 10 | 9 | 19
  No Diabetes | 44 | 40 | 84
Hypertension [Count of Participants; unit: Participants]
  Hypertension | 29 | 22 | 51
  No Hypertension | 25 | 27 | 52
Hyperlipidemia [Count of Participants; unit: Participants]
  Dyslipidemia | 33 | 26 | 59
  No Dylsipidemia | 21 | 23 | 44
Current Smoker [Count of Participants; unit: Participants]
  Yes | 28 | 30 | 58
  No | 26 | 18 | 44
  Unknown | 0 | 1 | 1
History of Stroke [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 53 | 49 | 102
Family History of Myocardial Infarction [Count of Participants; unit: Participants]
  Yes | 18 | 23 | 41
  No | 36 | 26 | 62
Infarct related artery [Count of Participants; unit: Participants]
  LCx | 4 | 3 | 7
  LAD | 22 | 17 | 39
  RCA | 25 | 28 | 53
  Multiple Arteries | 3 | 1 | 4
Ejection Fraction [Mean (Standard Deviation); unit: Percent of blood ejected] | 50.3 (10.0) | 50.1 (10.1) | 50.2 (10.0)
Ischemic Duration [Median (Inter-Quartile Range); unit: Minutes] | 144 [112 to 207] | 158 [115 to 214] | 146 [112 to 211]

OUTCOME MEASURES:

1. Primary Outcome: Infarct Size on Baseline Cardiac Magnetic Resonance Imaging (cMRI)
Description: Infarct size was quantified by delayed, contrast-enhanced MRI
Time Frame: Day 3-5 post-PCI
Population: There were 12 patients whose MRI data were not usable, including 6 in the post conditioning + PCI group and 6 in the standard PCI group.
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 47 | 43
ml | 20.1 [12.8 to 30.2] | 21.0 [13.8 to 30.6]
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 0.90, Kruskal-Wallis

2. Primary Outcome: Myocardial Salvage Index (MSI) on Baseline cMRI
Description: The myocardial salvage index (MSI) was calculated using the formula: MSI = (AAR - Infarct size) / AAR X 100 % where quantitative estimation of myocardium at risk (AAR) was measured as the hyperintense region on T2- weighted imaging. Measurements were performed using the QMass software package (Medis mc, Raleigh NC) by a single investigator who was blinded to treatment. The endocardial and epicardial borders were manually identified and the regions of interest (edema or scar) were automated as 2 standard deviations above the mean density of the myocardium.
Time Frame: Day 3-5 post-PCI
Population: There were 18 patients we were unable to obtain myocardial salvage indexes for, including 10 in the post conditioning + PCI group and 8 in the standard PCI group.
Measure: Median (Inter-Quartile Range); unit: (%)
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 43 | 41
(%) | 32.6 [20.6 to 49.7] | 32.7 [22.2 to 46.4]
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 0.81, Kruskal-Wallis

3. Primary Outcome: Micro Vascular Obstruction (MVO) on Baseline cMRI
Description: High T1 imaging was utilized for the determination of the presence or absence of MVO.
Time Frame: Day 3-5 post-PCI
Population: There were 8 patients in which were unable to determine the presence or absence of MVO, including 4 in the post conditioning + PCI group and 4 in the standard PCI group.
Measure: Count of Participants; unit: Participants
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 49 | 45
Participants | 31 | 25
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 0.45, Chi-squared

4. Secondary Outcome: Global Left Ventricular Ejection Fraction
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 54 | 49
Percent | 55.1 (10.8) | 54.0 (9.5)
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 0.58, t-test, 2 sided

5. Secondary Outcome: Infarct Size by Peak Troponin
Time Frame: over first 72 hour post PCI
Population: There were 31 patients who did not have a troponin drawn within the specified study protocol window, including 10 in the post conditioning + PCI group and 21 in the standard PCI group.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 43 | 28
ng/ml | 19.63 [3.55 to 72.36] | 14.44 [9.05 to 38.53]
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 0.86, Kruskal-Wallis

6. Secondary Outcome: Infarct Size by Peak Creatine Kinase (CK)
Time Frame: over first 72 hours post PCI
Population: There was 1 patient who did not have a CK lab test done in the standard PCI group.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 53 | 48
IU/L | 1701 [873 to 2854] | 1619 [801 to 2899]
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 1.00, Kruskal-Wallis

7. Secondary Outcome: Left Ventricular Remodeling (Left Ventricular End Diastolic Volume - LVEDV) as Measured by cMRl
Description: LVEDV was defined as the volume of blood in the left ventricle at end load or filling in diastole or the amount of blood in the ventricles just before systole.
Time Frame: baseline
Population: There were 4 patients who did not have an LVEDV measurement done, including 2 in the post conditioning + PCI group and 2 in the standard PCI group.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 51 | 47
mL | 149 [138 to 172] | 147 [133 to 170]
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 0.58, Kruskal-Wallis

8. Secondary Outcome: Left Ventricular Remodeling (Left Ventricular End Systolic Volume - LVESV) as Measured by cMRl
Description: LVESV was defined as the volume of blood in the left ventricle at the end of contraction, or systole, and the beginning of filling, or diastole.
Time Frame: baseline
Population: There were 4 patients who did not have an LVESV measurement done, including 2 in the post conditioning + PCI group and 2 in the standard PCI group.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Post Conditioning + PCI | Standard PCI
Number analyzed (Participants) | 51 | 47
mL | 70 [51 to 81] | 65 [55 to 86]
Statistical Analysis 1: Comparison: Post Conditioning + PCI vs Standard PCI; Test type: Superiority; p = 0.77, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | Post Conditioning + PCI | Standard PCI
All-Cause Mortality (participants affected / at risk) | 0/54 | 1/49
Serious Adverse Events (participants affected / at risk) | 2/54 | 2/49
Other Adverse Events (participants affected / at risk) | 13/54 | 7/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Conditioning + PCI (N=54) | Standard PCI (N=49)
CVA (Cardiac disorders) | 0 (0) | 1 (1)
Acute Stent Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization readmission for Heart Failure (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Conditioning + PCI (N=54) | Standard PCI (N=49)
Atriall Fibrillation/Flutter (Cardiac disorders) | 2 (2) | 2 (2)
Chest Pain (Cardiac disorders) | 1 (1) | 2 (2)
Groin hematoma (Vascular disorders) | 2 (2) | 3 (3)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
NSVT (Cardiac disorders) | 3 (4) | 0 (0)
VF/VT (Cardiac disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No